CLINICAL TRIAL: NCT06148324
Title: Promoting Wellness in Individuals With Traumatic Brain Injury: A Randomized Trial Assessing the Effectiveness of the Mindfulness, Exercise, Nutrition to Optimize Resilience (MENTOR) Program
Brief Title: MENTOR Wellness Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-00826
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; TBI; brain injury; wellness; physical activity; nutrition; chronic; mindfulness
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries; Motor Activity; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate treatment (IT) (Experimental): Participants randomized to the IT arm will receive the 8-week MENTOR program, followed by an 8-week retention period.
  Interventions: Behavioral: MENTOR Program
- Delayed treatment (DT) (Experimental): Participants randomized to the DT arm will have an 8-week waitlist period prior to starting the 8-week MENTOR program, followed by an 8-week retention period.
  Interventions: Behavioral: MENTOR Program

INTERVENTIONS:
Behavioral: MENTOR Program — MENTOR is an online wellness program covering 11 wellness modules: Exercise; Nutrition; Mindfulness; Spiritual Practice; Self-Care; Arts & Leisure; Rest & Relaxation; Outdoors in Nature; Relationships; Core Values; and Contribution to Others.
  The 8-week cycle comprises 40 hours of online group-based instruction and discussion, meeting up to five times per week.

SUMMARY:
This randomized trial aims to determine the effectiveness a virtual wellness intervention program in individuals with traumatic brain injury (TBI). Participants will be randomized at enrollment into two groups: immediate treatment (IT) and delayed treatment (DT) group. This study will also provide insights into the impact of these intervention's components in helping emotional, physical, and nutritional outcomes post-injury in the context of social determinants of health (SDOH).

ELIGIBILITY:
Inclusion Criteria:

* Have a medically-documented (e.g., EMS report, hospital record, physician record) or per medical monitor review complicated-mild, moderate, or severe TBI requiring admission to an acute inpatient rehabilitation unit
* Be at least 12 months post-TBI
* Have access to the internet on a computer, tablet, and/or smartphone.
* Speak and understand English or Spanish
* Agree to participate
* Are medically cleared by their primary physician, physiatrist, neurologist, rehabilitation therapist, or other recognized health professional to participate in the study

Exclusion Criteria:

* No history of complicated-mild, moderate, or severe TBI
* Less than 12 months post-TBI
* In minimally conscious or vegetative state
* Beginning a new treatment regimen (e.g., physical therapy, occupational therapy, vestibular therapy, psychotherapy, and/or medication) at study start that can influence study findings in the judgment of the principal investigator and/or medical monitor (participants whose treatment regimens are stable will be eligible)
* In the judgment of the principal investigator, medical monitor, and/or study team member, presence of significant cognitive impairment (i.e. delirium or dementia) sufficient to preclude meaningful informed consent and/or data collection
* In the judgment of the principal investigator, medical monitor, and/or study team member, significant or major disabling medical condition sufficient to preclude meaningful informed consent and/or data collection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Freiburg Mindfulness Inventory (FMI) Score at Baseline | Baseline
  14-item scale measuring mindfulness. Items are rated on a scale from 1 (rarely) to 4 (almost always); the total score is the sum of responses and ranges from 14 to 56; higher scores indicate greater levels of mindfulness.
Freiburg Mindfulness Inventory (FMI) Score at Post-Intervention Assessment | Post-Intervention Assessment (Week 8 for IT; Week 16 for DT)
  14-item scale measuring mindfulness. Items are rated on a scale from 1 (rarely) to 4 (almost always); the total score is the sum of responses and ranges from 14 to 56; higher scores indicate greater levels of mindfulness.
International Physical Activity Questionnaire (IPAQ) Score at Baseline | Baseline
  The IPAQ calculates the metabolic equivalent (MET) score by asking participants the days and minutes exercised in three categories of intensity (vigorous, moderate, and walking) during the previous one week. The following formula is used to calculate the MET: MET=8(vigorous activity) (minutes) + 4 (moderate activity)(minutes) +3.3 (walking activity) (minutes).
International Physical Activity Questionnaire Score at Post-Intervention Assessment | Post-Intervention Assessment (Week 8 for IT; Week 16 for DT)
  The IPAQ calculates the metabolic equivalent (MET) score by asking participants the days and minutes exercised in three categories of intensity (vigorous, moderate, and walking) during the previous one week. The following formula is used to calculate the MET: MET=8(vigorous activity) (minutes) + 4 (moderate activity)(minutes) +3.3 (walking activity) (minutes).
Health Promoting Lifestyle Profile II (HPLP-II) Score at Baseline | Baseline
  53-item self-assessment of nutritional and health-related habits. Items are rated on a scale from 1 (never) to 4 (routinely); the total score is the sum of responses and ranges from 52 to 208. Higher scores indicate nutritional and health-related habits that are more closely associated with good health outcomes.
Health Promoting Lifestyle Profile II (HPLP-II) Score at Post-Intervention Assessment | Post-Intervention Assessment (Week 8 for IT; Week 16 for DT)
  53-item self-assessment of nutritional and health-related habits. Items are rated on a scale from 1 (never) to 4 (routinely); the total score is the sum of responses and ranges from 52 to 208. Higher scores indicate nutritional and health-related habits that are more closely associated with good health outcomes.
Connor-Davidson Resilience Scale 10 (CD-RISC-10) Score at Baseline | Baseline
  10-item assessment of how participants feel when faced with various difficult situations. Each item is rated on a scale from 0 (not true at all) to (true nearly all the time). The total score is the sum of responses and ranges from 0 to 40; higher scores indicate greater resilience.
Connor-Davidson Resilience Scale 10 (CD-RISC-10) Score at Post-Retention Assessment | Post-Retention Period Assessment (Week 16 for IT; Week 24 for DT)
  10-item assessment of how participants feel when faced with various difficult situations. Each item is rated on a scale from 0 (not true at all) to (true nearly all the time). The total score is the sum of responses and ranges from 0 to 40; higher scores indicate greater resilience.
Perceived Stress Scale (PSS) Score at Baseline | Baseline
  10-item assessment of perceived stress. Each item is rated on a scale from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0 to 40; higher scores indicate higher perceived stress.
Perceived Stress Scale (PSS) Score at Post-Retention Assessment | Post-Retention Period Assessment (Week 16 for IT; Week 24 for DT)
  10-item assessment of perceived stress. Each item is rated on a scale from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0 to 40; higher scores indicate higher perceived stress.
Participation Assessment with Recombined Tools - Objective (PART-O) Score at Baseline | Baseline
  10-item assessment of participation in the community. Each item is rated on a scale from 0-5; the total score is the sum of responses and ranges from 0 to 50; higher scores indicate greater community participation.
Participation Assessment with Recombined Tools - Objective (PART-O) Score at Post-Retention Assessment | Post-Retention Period Assessment (Week 16 for IT; Week 24 for DT)
  10-item assessment of participation in the community. Each item is rated on a scale from 0-5; the total score is the sum of responses and ranges from 0 to 50; higher scores indicate greater community participation.
Quality of Life after Brain Injury (QOLIBRI) Score at Baseline | Baseline
  37-item assessment of quality of life following brain injury. Items rated on a scale from 1 (not at all) to 5 (very). The total score is the sum of responses and ranges from 37 to 185; higher scores indicate greater quality of life.
Quality of Life after Brain Injury (QOLIBRI) Score at Post-Retention Assessment | Post-Retention Period Assessment (Week 16 for IT; Week 24 for DT)
  37-item assessment of quality of life following brain injury. Items rated on a scale from 1 (not at all) to 5 (very). The total score is the sum of responses and ranges from 37 to 185; higher scores indicate greater quality of life.
12-Item Short Form Survey (SF-12) Score at Baseline | Baseline
  12-item assessment of general health. The raw score is the sum of responses; the raw score is transformed to a summary t-score with a mean of 50 and standard deviation of 10; higher scores indicate greater overall health.
12-Item Short Form Survey (SF-12) Score at Post-Retention Assessment | Post-Retention Period Assessment (Week 16 for IT; Week 24 for DT)
  12-item assessment of general health. The raw score is the sum of responses; the raw score is transformed to a summary t-score with a mean of 50 and standard deviation of 10; higher scores indicate greater overall health.
WHO-Quality of Life - Spirituality, Religious and Personal Beliefs module (WHOQOL-SRPB BREF) Score at Baseline | Baseline
  32-item assessment of how beliefs have affected different aspects of a participant's quality of life over the past two weeks. Items are rated on a scale from 1 (not at all) to 5 (an extreme amount). The total score is the sum of responses and ranges from 32 to 160; higher scores indicate beliefs have a greater impact on the participant's quality of life.
WHO-Quality of Life - Spirituality, Religious and Personal Beliefs module (WHOQOL-SRPB BREF) Score at Post-Retention Assessment | Post-Retention Period Assessment (Week 16 for IT; Week 24 for DT)
  32-item assessment of how beliefs have affected different aspects of a participant's quality of life over the past two weeks. Items are rated on a scale from 1 (not at all) to 5 (an extreme amount). The total score is the sum of responses and ranges from 32 to 160; higher scores indicate beliefs have a greater impact on the participant's quality of life.
Flourishing Scale Score at Baseline | Baseline
  8-item assessment of general prosperity. Each item is rated on a scale from 1 (strongly disagree) to 7 (strongly agree). The total score is the sum of responses and ranges from 8-56; higher scores indicate greater prosperity.
Flourishing Scale Score at Post-Retention Assessment | Post-Retention Period Assessment (Week 16 for IT; Week 24 for DT)
  8-item assessment of general prosperity. Each item is rated on a scale from 1 (strongly disagree) to 7 (strongly agree). The total score is the sum of responses and ranges from 8-56; higher scores indicate greater prosperity.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Bushnik, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared with researchers who provide a methodologically sound proposal to achieve aims in the approved protocol. The request may be submitted beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the researchers execute a data use agreement with NYU Langone Health. Requests may be directed to: Tamara.Bushnik@nyulangone.org. After 36 months, the data will be available in NYU Langone's data warehouse but without investigator support other than deposited metadata. Information regarding submitting requests and accessing data may be found at ICPSR Data Excellence Research Impact (umich.edu). The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Requests should be directed to Tamara.Bushnik@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. Proposals may be submitted up to 36 months following article publication. After 36 months, the data will be available in NYU Langone's data warehouse but without investigator support other than deposited metadata. Information regarding submitting requests and accessing data may be found at ICPSR Data Excellence Research Impact (umich.edu).